CLINICAL TRIAL: NCT01328041
Title: A Phase III Study to Demonstrate the Antiviral Activity and Safety of Dolutegravir in HIV-1 Infected Adult Subjects With Treatment Failure on an Integrase Inhibitor Containing Regimen.
Brief Title: A Study to Assess Dolutegravir in HIV-infected Subjects With Treatment Failure on an Integrase Inhibitor Containing Regimen.
Acronym: VIKING-3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: Shionogi (Industry); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 112574
Record Dates: First submitted 2011-03-31; First posted 2011-04-04 (Estimated); Results first posted 2014-07-21 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2015-12

CONDITIONS: Infection, Human Immunodeficiency Virus
Keywords: GSK1349572; resistance to raltegravir or elvitegravir; Integrase inhibitor; ART-experienced; dolutegravir
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome | interventions — dolutegravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- dolutegravir (Experimental): dolutegravir plus background antiretroviral therapy optimised at Day 8
  Interventions: Drug: dolutegravir

INTERVENTIONS:
Drug: dolutegravir — 50 mg twice daily

SUMMARY:
The purpose of this trial is to assess the antiviral activity and safety of a dolutegravir (DTG) containing regimen in HIV-1 infected, antiretroviral therapy (ART)-experienced adults with current or historical failure on an integrase inhibitor (INI) containing regimen. The study will assess DTG 50mg twice daily administered initially with the current failing ART regimen but then with an optimised background ART regimen (OBR) after Day 7. The first analyses will be conducted after the last subject enrolled has completed 24 weeks. Subjects may remain on study after Week 24.

DETAILED DESCRIPTION:
ING112574 is a Phase 3, multicentre, open-label, single arm study to assess the antiviral activity and safety of DTG containing regimen in HIV-1 infected ART-experienced adults with historical or current evidence of resistance to RAL or ELV. Initially, a minimum of 100 subjects will be enrolled to receive DTG 50mg twice daily with the current failing regimen for 7 days but with OBR from Day 8. Subjects must also have documented genotypic and/or phenotypic resistance to at least one compound in two or more of the other approved classes of ART but must also be able to include at least one fully active drug in the OBR to be started Day 8. The first data cut will take place after the (approximate) 100th subject enrolled completes the Week 24 visit. Enrollment will continue until a further 50 to 100 subjects have been recruited. All subjects who successfully complete 24 weeks of treatment will continue to have access to DTG until it is locally available as long as they continue to derive clinical benefit.

ViiV Healthcare is the sponsor of this study.

ELIGIBILITY:
Inclusion Criteria:

* Screening plasma HIV-1 RNA ≥500 copies/mL
* ART-experienced, INI-experienced, DTG naïve
* Experienced virological failure on raltegravir (RAL) or elvitegravir (ELV) regimen
* The subject's HIV-1 shows resistance to RAL or ELV at Screening or at prior time point of virological failure on RAL or ELV
* Documented resistance to at least one drug from each of three or more of all approved classes of ART
* Be able to receive at least one fully active drug as part of the OBR from Day 8
* Women capable of becoming pregnant must use appropriate contraception during the study (as defined by the protocol)
* Willing and able to understand and provide signed and dated written informed consent prior to Screening.

Exclusion Criteria:

* Women who are pregnant or breast feeding
* An active AIDS-defining condition at Screening (except cutaneous Kaposi's sarcoma not requiring systemic therapy or CD4+ <200c/mm3)
* Moderate to severe hepatic impairment as defined by Child-Pugh classification
* Anticipated need for HCV therapy during the first 24 weeks of the study
* Recent history of any upper or lower gastrointestinal bleed, with the exception of anal or rectal bleeding
* Allergy or intolerance to the study drugs or their components or drugs of their class
* Malignancy within the past 6 months
* Treatment with an HIV-1 therapeutic vaccine within 90 days of Screening
* Treatment with radiation therapy, cytotoxic chemotherapeutic agents or any immunomodulator within 28 days of Screening
* Treatment with any agent, other than licensed ART, with documented activity against HIV-1 in vitro within 28 days of first dose of investigational product
* Treatment with etravirine, efavirenz, or nevirapine within 14 days of Day 1(etravirine may be used if coadministered with lopinivir/ritonavir or darunavir/ritonavir)
* Treatment with tipranivir/ritonavir, fosamprenavir, or fosamprenavir/ritonavir within 28 days prior to Screening
* Verified Grade 4 laboratory abnormality at Screening
* ALT> 5 times the upper limit of normal (ULN) at Screening
* ALT ≥ 3X ULN and bilirubin > 1.5 X ULN (with 35% direct bilirubin) at Screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2011-05; Primary Completion 2012-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (65):
- United States (35):
  - GSK Investigational Site, Beverly Hills, California
  - GSK Investigational Site, Fountain Valley, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, New Haven, Connecticut
  - GSK Investigational Site, Norwalk, Connecticut
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Ft. Pierce, Florida
  - GSK Investigational Site, Miami Beach, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Lafayette, Louisiana
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Jackson, Mississippi
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Newark, New Jersey
  - GSK Investigational Site, Albany, New York
  - GSK Investigational Site, Buffalo, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Valhalla, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Toledo, Ohio
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Providence, Rhode Island
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Annandale, Virginia
  - GSK Investigational Site, Seattle, Washington
- Belgium (2):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Liège
- Canada (4):
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
- France (9):
  - GSK Investigational Site, Aulnay-sous-Bois
  - GSK Investigational Site, Bobigny
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Garches
  - GSK Investigational Site, Gonesse
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Nice
  - GSK Investigational Site, Orléans
  - GSK Investigational Site, Paris
- Italy (6):
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Bergamo, Lombardy
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Turin, Piedmont
  - GSK Investigational Site, Bagno A Ripoli (FI), Tuscany
  - GSK Investigational Site, Florence, Tuscany
- Portugal (3):
  - GSK Investigational Site, Amadora
  - GSK Investigational Site, Coimbra
  - GSK Investigational Site, Lisbon
- Spain (6):
  - GSK Investigational Site, A Coruña
  - GSK Investigational Site, Alicante
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Seville

REFERENCES:
- [Background] Eron JJ, Clotet B, Durant J, Katlama C, Kumar P, Lazzarin A, Poizot-Martin I, Richmond G, Soriano V, Ait-Khaled M, Fujiwara T, Huang J, Min S, Vavro C, Yeo J; VIKING Study Group. Safety and efficacy of dolutegravir in treatment-experienced subjects with raltegravir-resistant HIV type 1 infection: 24-week results of the VIKING Study. J Infect Dis. 2013 Mar 1;207(5):740-8. doi: 10.1093/infdis/jis750. Epub 2012 Dec 7. PMID 23225901
- [Derived] Castagna A, Maggiolo F, Penco G, Wright D, Mills A, Grossberg R, Molina JM, Chas J, Durant J, Moreno S, Doroana M, Ait-Khaled M, Huang J, Min S, Song I, Vavro C, Nichols G, Yeo JM; VIKING-3 Study Group. Dolutegravir in antiretroviral-experienced patients with raltegravir- and/or elvitegravir-resistant HIV-1: 24-week results of the phase III VIKING-3 study. J Infect Dis. 2014 Aug 1;210(3):354-62. doi: 10.1093/infdis/jiu051. Epub 2014 Jan 19. PMID 24446523

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants (par.) having documented Human immunodeficiency virus type 1 (HIV-1) infection with a plasma HIV-1 Ribonucleic acid(RNA) >=500 copies per milliliter (c/mL) at Screening, Antiretroviral therapy (ART)-experienced and on stable ART for at least one month prior to Screening were enrolled
Pre-assignment Details: A total of 139 par. were screen failures and 183 par. entered the single arm, open-label study.
Groups:
- Dolutegravir 50 mg BID: Participants received dolutegravir (DTG) 50 milligrams (mg) twice a day (BID).
Period: Overall Study
Arm/Group | Dolutegravir 50 mg BID
Started | 183
Completed | 126
Not Completed | 57
Not completed — Adverse Event | 7
Not completed — Lack of Efficacy | 27
Not completed — Protocol Violation | 7
Not completed — Lost to Follow-up | 7
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 7

BASELINE CHARACTERISTICS:
Groups:
- Dolutegravir 50 mg BID: Participants received DTG 50 mg BID.
Arm/Group | Dolutegravir 50 mg BID
Number analyzed (Participants) | 183
Age, Continuous [Median (Full Range); unit: Years] | 48 [19 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 141
Race/Ethnicity, Customized [Number; unit: participants]
  African American/African Heritage | 49
  American Indian or Alaska Native and White | 1
  Asian-Central/South Asian Heritage | 1
  White | 130
  White and African American/African Heritage | 2

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Plasma HIV-1 RNA at Day 8
Description: Mean change from Baseline in Plasma Human Immunodeficiency Virus-1 (HIV-1) Ribonucleic Acid (RNA) at Day 8 was calculated as the Day 8 value minus the Baseline value. The last observation was carried forward if a participant had missed the Day 8 visit. The Baseline observation was carried forward if a participant had discontinued the treatment before Day 8. Blood samples for assessment of HIV-1 RNA levels were collected at Baseline and Day 8.
Time Frame: Baseline and Day 8
Population: Intent-to-Treat-Exposed (ITT-E) Population: all participants who received at least one dose of study drug. Only participants who had Day 8 observations were considered for analysis.
Measure: Mean (Standard Deviation); unit: log10 copies/milliliter (mL)
Arm/Group | Dolutegravir 50 mg BID
Number analyzed (Participants) | 182
log10 copies/milliliter (mL) | -1.432 (0.6070)
Statistical Analysis 1: Comparison: Dolutegravir 50 mg BID; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — The P value was derived by the null hypothesis testing of no change from Baseline in HIV-1 RNA at Day 8 at the two-sided 5% significance level using a single sample t-test; T distribution = -1.432, 95% CI 2-sided [-1.520 to -1.343]

2. Primary Outcome: Number of Participants With HIV-1 RNA Less Than 50 Copies/mL at Week 24
Description: The number of participants who had viral load <50 copies/mL at Week 24 based on the Food and Drug Administration's Snapshot algorithm was assessed. This algorithm treats all participants without HIV-1 RNA data at the visit of interest (VOI [due to missing data/discontinuation of investigational product prior to the visit window]) as nonresponders, as well as participants who switched their concomitant antiretroviral (ART) prior to the VOI as follows: background ART substitutions not permitted per protocol; background ART substitutions permitted per protocol, however the decision to switch was not documented as being before or at the first on-treatment visit after switching to optimized background regimen (i.e., Week 4) where HIV-1 RNA was assessed. Otherwise, virologic success/failure was to be determined by the last available HIV-1 RNA assessment while the participant was on treatment within the VOI analysis window.
Time Frame: Week 24
Population: ITT-E Population
Measure: Number; unit: participants
Arm/Group | Dolutegravir 50 mg BID
Number analyzed (Participants) | 183
participants | 126
Statistical Analysis 1: Comparison: Dolutegravir 50 mg BID; Test type: Superiority or Other; percentage of participants = 69, 95% CI 2-sided [62 to 76] — The estimated value represents the percentage of participants with HIV-1 RNA less than 50 copies/mL at Week 24

3. Primary Outcome: Number of Participants With HIV-1 RNA Less Than 50 Copies/mL at Week 48
Description: The number of participants who had viral load <50 copies/mL at Week 48 based on the Food and Drug Administration's Snapshot algorithm was assessed. This algorithm treats all participants without HIV-1 RNA data at the visit of interest (VOI [due to missing data/discontinuation of investigational product prior to the visit window]) as nonresponders, as well as participants who switched their concomitant antiretroviral (ART) prior to the VOI as follows: background ART substitutions not permitted per protocol; background ART substitutions permitted per protocol, however the decision to switch was not documented as being before or at the first on-treatment visit after switching to optimized background regimen (i.e., Week 4) where HIV-1 RNA was assessed. Otherwise, virologic success/failure was to be determined by the last available HIV-1 RNA assessment while the participant was on treatment within the VOI analysis window.
Time Frame: Week 48
Population: ITT-E Population
Measure: Number; unit: participants
Arm/Group | Dolutegravir 50 mg BID
Number analyzed (Participants) | 183
participants | 116
Statistical Analysis 1: Comparison: Dolutegravir 50 mg BID; Test type: Superiority or Other; percentage of participants = 63, 95% CI 2-sided [56 to 70] — The estimated value represents the percentage of participants with HIV-1 RNA less than 50 copies/mL at Week 48

4. Primary Outcome: Number of Participants With Any Adverse Event (AE) or Any Serious Adverse Event (SAE)
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, or is an event of possible drug-induced liver injury.
Time Frame: From the day of the first dose of study drug until end of treatment visit for each participant, up to Week 180 (median of 758 days)
Population: Safety Population: all participants who received at least one dose of study drug
Measure: Number; unit: participants
Arm/Group | Dolutegravir 50 mg BID
Number analyzed (Participants) | 183
participants
  Any AE | 169
  Any SAE | 46

5. Primary Outcome: Number of Participants With Adverse Events of the Indicated Severity, Per the Division of Acquired Immune Deficiency Syndrome (DAIDS) Grading Scale
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, or is an event of possible drug-induced liver injury. AE/SAE severity was graded according to the DAIDS grading scale. The DAIDS displays events as Grades 1-4 based on this general guideline: Grade (G) 1, mild; G2, moderate; G3, severe; G4, potentially life threatening.
Time Frame: as for outcome 4
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Dolutegravir 50 mg BID
Number analyzed (Participants) | 183
participants
  Grade 1 | 45
  Grade 2 | 64
  Grade 3 | 44
  Grade 4 | 16

6. Primary Outcome: Number of Participants With the Maximum Post-Baseline-emergent Clinical Chemistry Toxicities of the Indicated Grade
Description: The severity of clinical chemistry toxicities was graded according to the DAIDS toxicity scale. The DAIDS displays events as Grades 1-5 based on this general guideline: Grade (G) 1, mild; G2, moderate; G3, severe; G4, life threatening; G5, death related to toxicity.
Time Frame: as for outcome 4
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Dolutegravir 50 mg BID
Number analyzed (Participants) | 183
participants
  Grade 1 | 49
  Grade 2 | 67
  Grade 3 | 43
  Grade 4 | 16

7. Primary Outcome: Number of Participants With the Maximum Post-Baseline-emergent Hematology Toxicities of the Indicated Grade
Description: The severity of hematology toxicities was graded according to the DAIDS. The DAIDS displays events as Grades 1-5 based on this general guideline: Grade (G) 1, mild; G2, moderate; G3, severe; G4, life threatening; G5, death related to toxicity.
Time Frame: as for outcome 4
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Dolutegravir 50 mg BID
Number analyzed (Participants) | 183
Participants
  Grade 1 | 31
  Grade 2 | 15
  Grade 3 | 4
  Grade 4 | 2

8. Secondary Outcome: Number of Participants With Plasma HIV-1 RNA Less Than 400 and 50 Copies/mL at Baseline; Day 8; and Weeks 4, 8, 12, 16, 24, 32, 40, and 48
Description: The number of participants with plasma HIV-1 RNA less than 400 and 50 copies (c)/mL at Baseline; Day 8; and Weeks 4, 8, 12, 16, 24, 32, 40 and 48 based on the Food and Drug Administration's Snapshot algorithm was assessed. This algorithm treats all participants without HIV-1 RNA data at the visit of interest (VOI [due to missing data/discontinuation of investigational product prior to the visit window]) as nonresponders, as well as participants who switched their concomitant antiretroviral (ART) prior to the VOI as follows: background ART substitutions not permitted per protocol; background ART substitutions permitted per protocol, however the decision to switch was not documented as being before or at the first on-treatment visit after switching to optimized background regimen (i.e., Week 4) where HIV-1 RNA was assessed. Otherwise, virologic success/failure was to be determined by the last available HIV-1 RNA assessment while the par. was on treatment within the VOI analysis window
Time Frame: Baseline; Day 8; and Weeks 4, 8, 12, 16, 24, 32, 40, and 48
Population: ITT-E Population
Measure: Number; unit: participants
Arm/Group | Dolutegravir 50 mg BID
Number analyzed (Participants) | 183
participants
  HIV-1 RNA <50 c/mL, Baseline | 1
  HIV-1 RNA <50 c/mL, Day 8 | 28
  HIV-1 RNA <50 c/mL, Week 4 | 98
  HIV-1 RNA <50 c/mL, Week 8 | 112
  HIV-1 RNA <50 c/mL, Week 12 | 116
  HIV-1 RNA <50 c/mL, Week 16 | 116
  HIV-1 RNA <50 c/mL, Week 24 | 126
  HIV-1 RNA <50 c/mL, Week 32 | 117
  HIV-1 RNA <50 c/mL, Week 40 | 108
  HIV-1 RNA <50 c/mL, Week 48 | 116
  HIV-1 RNA <400 c/mL, Baseline | 8
  HIV-1 RNA <400 c/mL, Day 8 | 82
  HIV-1 RNA <400 c/mL, Week 4 | 145
  HIV-1 RNA <400 c/mL, Week 8 | 146
  HIV-1 RNA <400 c/mL, Week 12 | 142
  HIV-1 RNA <400 c/mL, Week 16 | 139
  HIV-1 RNA <400 c/mL, Week 24 | 135
  HIV-1 RNA <400 c/mL, Week 32 | 127
  HIV-1 RNA <400 c/mL, Week 40 | 119
  HIV-1 RNA <400 c/mL, Week 48 | 125

9. Secondary Outcome: Number of Participants With Plasma HIV-1 RNA Less Than 400 and 50 Copies/mL From Week 48 Every 12 Weeks up to Study Completion
Description: The number of participants with plasma HIV-1 RNA less than 400 and 50 copies (c)/mL was assessed at Weeks 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, 168 and 180 using data of observed cases. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: From Week 48 every 12 weeks up to study completion.
Population: ITT-E Population
Measure: Number; unit: Participants
Arm/Group | Dolutegravir 50 mg BID
Number analyzed (Participants) | 183
Participants
  HIV-1 RNA <50 c/mL, Week 48, n =146 | 121 [40.0 to 330.0]
  HIV-1 RNA <50 c/mL, Week 60, n=142 | 110 [60.0 to 350.0]
  HIV-1 RNA <50 c/mL, Week 72, n=138 | 116 [80.0 to 350.0]
  HIV-1 RNA <50 c/mL, Week 84, n=138 | 108 [100.0 to 350.0]
  HIV-1 RNA <50 c/mL, Week 96, n=120 | 101 [110.0 to 360.0]
  HIV-1 RNA <50 c/mL, Week 108, n=98 | 81 [130.0 to 400.0]
  HIV-1 RNA <50 c/mL, Week 120, n=82 | 72 [130.0 to 420.0]
  HIV-1 RNA <50 c/mL, Week 132, n=61 | 49 [170.0 to 440.0]
  HIV-1 RNA <50 c/mL, Week 144, n=45 | 37 [200.0 to 440.0]
  HIV-1 RNA <50 c/mL, Week 156, n=32 | 28 [200.0 to 450.0]
  HIV-1 RNA <50 c/mL, Week 168, n=24 | 20 [540.0 to 1220.0]
  HIV-1 RNA <50 c/mL, Week 180, n=6 | 4 [655.0 to 1405.0]
  HIV-1 RNA <400 c/mL, Week 48, n=146 | 134 [730.0 to 1460.0]
  HIV-1 RNA <400 c/mL, Week 60, n=142 | 131 [690.0 to 1460.0]
  HIV-1 RNA <400 c/mL, Week 72, n=138 | 130 [720.0 to 1380.0]
  HIV-1 RNA <400 c/mL, Week 84, n=138 | 127
  HIV-1 RNA <400 c/mL, Week 96, n=120 | 111
  HIV-1 RNA <400 c/mL, Week 108, n=98 | 92
  HIV-1 RNA <400 c/mL, Week 120, n=82 | 80
  HIV-1 RNA <400 c/mL, Week 132, n=61 | 59
  HIV-1 RNA <400 c/mL, Week 144, n=45 | 44
  HIV-1 RNA <400 c/mL, Week 156, n=32 | 31
  HIV-1 RNA <400 c/mL, Week 168, n=24 | 23
  HIV-1 RNA <400 c/mL, Week 180, n=6 | 5

10. Secondary Outcome: Mean Change From Baseline in Plasma HIV-1 RNA at Day 8 and Weeks 4, 8, 12, 16, 24, 32, 40, and From Week 48 Every 12 Weeks up to Study Completion
Description: Mean change from Baseline in plasma HIV-1 RNA was assesseed at Day 8 and Weeks 4, 8, 12, 16, 24, 32, 40, 48 , 60, 72, 84, 96, 108, 120, 132, 144, 156, 168, and 180 using data of the observed cases. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Day 8; Weeks 4, 8, 12, 16, 24, 32, 40, and From Week 48 Every 12 Weeks up to Study completion (Up to Week 180)
Population: ITT-E Population. Only those participants with data available at the indicated time points were considered for analysis (represented by n=X in the category titles). Different participants may have been analyzed at different time points, so the overall number of participants analyzed reflects everyone in the ITT-E Population.
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Dolutegravir 50 mg BID
Number analyzed (Participants) | 183
Log10 copies/mL
  Day 8, n=182 | -1.432 (0.607) [0.0 to 60.0]
  Week 4, n=180 | -2.088 (0.885) [0.0 to 71.0]
  Week 8, n=179 | -2.101 (0.987) [0.0 to 81.0]
  Week 12, n=174 | -2.113 (1.069) [0.0 to 100.0]
  Week 16, n=165 | -2.216 (1.005) [20.0 to 130.0]
  Week 24, n=164 | -2.211 (1.023) [20.0 to 130.0]
  Week 32, n=146 | -2.373 (0.926) [20.0 to 160.0]
  Week 40, n=144 | -2.301 (0.955) [30.0 to 180.0]
  Week 48, n=146 | -2.321 (0.981) [40.0 to 190.0]
  Week 60, n=142 | -2.356 (0.928) [50.0 to 210.0]
  Week 72, n=138 | -2.390 (0.941)
  Week 84, n=138 | -2.311 (0.996) [80.0 to 240.0]
  Week 96, n=120 | -2.346 (1.008) [80.0 to 270.0]
  Week 108, n=98 | -2.394 (0.966) [80.0 to 280.0]
  Week 120, n=82 | -2.515 (0.904) [100.0 to 280.0]
  Week 132, n=61 | -2.456 (0.988) [100.0 to 320.0]
  Week 144, n=45 | -2.585 (0.983) [130.0 to 350.0]
  Week 156, n=32 | -2.595 (1.009) [155.0 to 345.0]
  Week 168, n=24 | -2.719 (0.898) [155.0 to 380.0]
  Week 180, n=6 | -2.425 (1.557) [140.0 to 230.0]

11. Secondary Outcome: Absolute Values for CD4+ Cell Counts at Baseline, Day 8 and Weeks 4, 8, 12, 16, 24, 32, 40, and 48 and for CD8+ Cell Counts at Baseline and Weeks 4, 12, 24, and 48
Description: Absolute values for CD4+ cell counts were assessed at Baseline, Day 8 and Weeks 4, 8, 12, 16, and 24, and absolute values for CD8+ cell counts were assessed at Baseline and Weeks 4, 12, 24, and 48.
Time Frame: Baseline, Day 8 and Weeks 4, 8, 12, 16, 24, 32, 40, and 48
Population: as for outcome 10
Measure: Median (Inter-Quartile Range); unit: Cells per millimeters cubed (cells/mm^3)
Arm/Group | Dolutegravir 50 mg BID
Number analyzed (Participants) | 183
Cells per millimeters cubed (cells/mm^3)
  CD4+, Baseline, n=183 | 140.0 (0.607) [40.0 to 330.0]
  CD4+, Day 8, n=181 | 170.0 (0.885) [60.0 to 350.0]
  CD4+, Week 4, n=178 | 185.0 (0.987) [80.0 to 350.0]
  CD4+, Week 8, n=178 | 210.0 (1.069) [100.0 to 350.0]
  CD4+, Week 12, n=171 | 210.0 (1.005) [110.0 to 360.0]
  CD4+, Week 16, n=165 | 210.0 (1.023) [130.0 to 400.0]
  CD4+, Week 24, n=163 | 250.0 (0.926) [130.0 to 420.0]
  CD4+, Week 32, n=147 | 270.0 (0.955) [170.0 to 440.0]
  CD4+, Week 40, n=143 | 290.0 (0.981) [200.0 to 440.0]
  CD4+, Week 48, n=145 | 310.0 (0.928) [200.0 to 450.0]
  CD8+, Week 4, n=181 | 860.0 (0.941) [540.0 to 1220.0]
  CD8+, Week 4, n=176 | 970.0 (0.996) [655.0 to 1405.0]
  CD8+, Week 12, n=170 | 1015.0 (1.008) [730.0 to 1460.0]
  CD8+, Week 24, n=154 | 1020.0 (0.966) [690.0 to 1460.0]
  CD8+, Week 48, n=140 | 1000.0 (0.904) [720.0 to 1380.0]

12. Secondary Outcome: Median Change From Baseline in CD4+ Cell Counts at Day 8 and Weeks 4, 8, 12, 16, 24, 32, 40, and From Week 48 Every 12 Weeks Until Study Completion
Description: Median change from Baseline in CD4+ cell counts was assessed at Day 8 and Weeks 4, 8, 12, 16, 24, 32, 40, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, 168, and 180. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Day 8; Weeks 4, 8, 12, 16, 24, 32, 40, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, 168 and 180. v
Population: as for outcome 10
Measure: Median (Inter-Quartile Range); unit: Cells per millimeters cubed (cells/mm^3)
Arm/Group | Dolutegravir 50 mg BID
Number analyzed (Participants) | 183
Cells per millimeters cubed (cells/mm^3)
  CD4+, Day 8, n=181 | 20.0 [0.0 to 60.0]
  CD4+, Week 4, n=178 | 30.0 [0.0 to 71.0]
  CD4+, Week 8, n=178 | 40.0 [0.0 to 81.0]
  CD4+, Week 12, n=171 | 50.0 [0.0 to 100.0]
  CD4+, Week 16, n=165 | 60.0 [20.0 to 130.0]
  CD4+, Week 24, n=163 | 61.0 [20.0 to 130.0]
  CD4+, Week 32, n=147 | 100.0 [20.0 to 160.0]
  CD4+, Week 40, n=143 | 90.0 [30.0 to 180.0]
  CD4+, Week 48, n=145 | 110.0 [40.0 to 190.0]
  CD4+, Week 60, n=142 | 120.0 [50.0 to 210.0]
  CD4+, Week 72, n=138 | 140.0 [60.0 to 231.0]
  CD4+, Week 84, n=137 | 150.0 [80.0 to 240.0]
  CD4+, Week 96, n=117 | 160.0 [80.0 to 270.0]
  CD4+, Week 108, n=98 | 180.5 [80.0 to 280.0]
  CD4+, Week 120, n=82 | 180.0 [100.0 to 280.0]
  CD4+, Week 132, n=61 | 221.0 [100.0 to 320.0]
  CD4+, Week 144, n=46 | 205.0 [130.0 to 350.0]
  CD4+, Week 156, n=32 | 225.0 [155. to 345.0]
  CD4+, Week168, n=24 | 265.0 [155.0 to 380.0]
  CD4+, Week180, n=6 | 170.5 [140.0 to 230.0]

13. Secondary Outcome: Ratio of CD4+/CD8+ Cell Count at Baseline and Weeks 4, 12, 24, and 48
Description: The ratio of CD4+/CD8+ cell count (measured in cells/mm^3) was assessed at Baseline and at Weeks 4, 12, 24, and 48. The ratio was calculated as the CD4+ cell count divided by CD8+ cell count.
Time Frame: Baseline; Weeks 4, 12, 24, and 48
Population: as for outcome 10
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Dolutegravir 50 mg BID
Number analyzed (Participants) | 183
ratio
  Baseline, n=180 | 0.15 [0.05 to 0.34]
  Week 4, n=176 | 0.19 [0.09 to 0.37]
  Week 12, n=170 | 0.21 [0.10 to 0.46]
  Week 24, n=154 | 0.26 [0.14 to 0.46]
  Week 48, n=140 | 0.32 [0.19 to 0.52]

14. Secondary Outcome: Number of Participants With HIV-1 Disease Progression (Acquired Immune Deficiency Syndrome [AIDS] or Death)
Description: The number of participants with HIV-1 disease progression (AIDS or death) was assessed per the Centers for Disease Control and Prevention (CDC) 1993 revised classification system for HIV infection and expanded surveillance case definition for AIDS among adolescents and adults. The CDC classifies HIV infection as Category A (participants with asymptomatic HIV infection, acute HIV infection with accompanying illness, or persistent generalized lymphadenopathy), Category B (participants with symptomatic non-AIDS condition, i.e., conditions that are attributed to HIV infection or are indicative of a defect in cell-mediated immunity; or conditions are considered by physicians to have a clinical course or to require management that is complicated by HIV infection), and Category C (includes AIDS indicator conditions as defined by diagnostic or presumptive measures).
Time Frame: as for outcome 4
Population: ITT-E Population
Measure: Number; unit: Participants
Arm/Group | Dolutegravir 50 mg BID
Number analyzed (Participants) | 183
Participants
  Progression from CDC Class A to Class C Event | 1 [4.18 to 5.36]
  Progression from CDC Class B to Class C Event | 2 [2.15 to 3.15]
  Progression from CDC Class C to New Class C Event | 6
  Progression from Classes A, B, or C to Death | 2

15. Secondary Outcome: Cmax and Ctau of DTG
Description: The maximum plasma concentration (Cmax) and the concentration at the end of a dosing interval (Ctau) of DTG were assessed by a population pharmacokinetic (PK) modeling approach using pooled DTG PK data from multiple studies. For this study, blood samples for pharmacokinetic assessments were collected pre-dose on Day 8 and at Weeks 4 and 24, at 1-3 hours post-dose on Day 8, and at 1-3 hours or 4-12 hours post-dose at Weeks 4 and 24.
Time Frame: Day 8, Week 4, and Week 24
Population: The Pharmacokinetic (PK) Concentration Population: all subjects who received DTG, had undergone PK sampling during the study, and provided evaluable DTG plasma concentration data.
Measure: Geometric Mean (95% Confidence Interval); unit: Micrograms per milliliter (µg/mL)
Arm/Group | Dolutegravir 50 mg BID
Number analyzed (Participants) | 183
Micrograms per milliliter (µg/mL)
  Cmax | 4.74 [4.18 to 5.36]
  Ctau | 2.60 [2.15 to 3.15]

16. Secondary Outcome: AUC(0-tau) and AUC(0-24) of DTG
Description: The area under the time concentration curve over the dosing interval (AUC[0-tau]) and from 0 to 24 hours (AUC[0-24]) of DTG was assessed by a population PK modeling approach using pooled DTG PK data from multiple studies. For this study, blood samples for pharmacokinetic assessments were collected pre-dose on Day 8 and at Weeks 4 and 24, at 1-3 hours post-dose on Day 8, and at 1-3 hours or 4-12 hours post-dose at Weeks 4 and 24.
Time Frame: Day 8, Week 4, and Week 24
Population: as for outcome 15
Measure: Geometric Mean (95% Confidence Interval); unit: µg*hour/mL
Arm/Group | Dolutegravir 50 mg BID
Number analyzed (Participants) | 183
µg*hour/mL
  AUC(0-tau) | 36.7 (91) [35.0 to 38.6]
  AUC(0-24) | 73.5 (113) [70.0 to 77.1]

17. Secondary Outcome: C0 Assessment of DTG
Description: The plasma DTG concentration immediately prior to dosing at steady state (C0) was assessed at Day 8, Week 4, and Week 24. Blood samples for pharmacokinetic assessments were collected pre-dose and 1-3 hours post-dose on Day 8 and at Week 4 and 4-12 hours post-dose at Week 24. Different participants may have been analyzed at different time points, so the overall number of participants analyzed reflects everyone in the Pharmacokinetic Parameter Population.
Time Frame: Day 8, Week 4, and Week 24
Population: Pharmacokinetic (PK) Parameter Population: all participants who received DTG, underwent PK sampling during the study, and provided an evaluable estimate of C0. Only participants with data available at the indicated time points were considered for analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Dolutegravir 50 mg BID
Number analyzed (Participants) | 161
µg/mL
  Day 8, n=148 | 2.36 (91)
  Week 4, n=161 | 1.90 (113)
  Week 24, n=135 | 2.14 (93)

18. Secondary Outcome: Number of Participants With the Indicated Treatment-emergent Integrase (IN) Mutations Detected at the Time of Protocol-defined Virologic Failure (PDVF) as a Measure of Genotypic Resistance
Description: An analysis of changes at specific amino acids in the IN coding region associated with resistance to raltegravir, elvitegravir, or DTG was performed at Day 1 and at the time of PDVF. PDVF is a <0.5 log10 copies(c)/mL decrease in plasma HIV-1 RNA at Day 8 unless the absolute value is <400 c/mL. PDVF after Day 8 is defined as virological non-respones (decrease in plasma HIV-1 RNA of <1 log10 c/mL by Week 16, with subsequent confirmation, unless plasma HIV-1 RNA <400 c/mL and confirmed plasma HIV-1 RNA levels >=400 c/mL on or after Week 24) and virological rebound (confirmed rebound in plasma HIV-1 RNA levels to >=400 c/mL after prior confirmed suppression to <400 c/mL and confirmed plasma HIV-1 RNA levels >1 log10 c/mL above the nadir value [nadir: >=400 c/mL]).
Time Frame: as for outcome 4
Population: PDVF Genotypic Resistance Populations: all participants in the ITT-E Population with available on-treatment genotypic resistance data at the time of PDVF. Only participants with Baseline IN mutations with PDVF who had paired Baseline and time of PDVF samples were considered for analysis.
Measure: Number; unit: participants
Arm/Group | Dolutegravir 50 mg BID
Number analyzed (Participants) | 42
participants
  Any IN mutation | 25
  T97A | 8
  T97T/A | 4
  E138A | 1
  E138E/A | 1
  E138E/K | 3
  E138K | 4
  E138T/A | 1
  N155H | 6
  N155N/H | 1
  Q148H | 3
  Q148Q/H | 2
  Q148R | 1
  Q148Q/R/K | 1
  G140G/S | 1
  G140S | 3
  L74L/M/V | 1
  L74L/M | 1
  L74I | 1
  E92E/Q | 2
  S147G | 2
  E157E/Q | 1
  V151V/M/I | 1
  Y143Y/H | 1

19. Secondary Outcome: Number of Participants With the Indicated Fold Increase in DTG FC (Fold Change in IC50 Relative to Wild-type Virus) Between Baseline and the Time of PDVF, as a Measure of Post-Baseline Phenotypic Resistance
Description: The FC in IC50 (50% inhibitory concentration) for DTG relative to wild-type virus was determined for virus isolated at Baseline and at the time of PDVF. The number of participants with the indicated change (ratio) in the two values at the time of PDVF is presented. PDVF is defined as a <0.5 log10 copies/mL decrease in plasma HIV-1 RNA at Day 8 unless the absolute value is <400 copies/mL. PDVF after Day 8 was defined for virological non-response (decrease in plasma HIV-1 RNA of less than 1 log10 copies/mL by Week 16, with subsequent confirmation, unless plasma HIV-1 RNA <400 copies/mL and confirmed plasma HIV-1 RNA levels >=400 copies/mL on or after Week 24) and virological rebound (confirmed rebound in plasma HIV-1 RNA levels to >=400 copies/mL after prior confirmed suppression to <400 copies/mL and confirmed plasma HIV-1 RNA levels >1 log10 copies/mL above the nadir value, where nadir is >=400 copies/mL).
Time Frame: as for outcome 4
Population: PDVF Phenotypic Resistance Populations. Only participants with Baseline DTG IC50 with PDVF who had paired Baseline and time of virological failure samples were considered for analysis.
Measure: Number; unit: Participants
Arm/Group | Dolutegravir 50 mg BID
Number analyzed (Participants) | 45
Participants
  <1 fold | 6
  1-<2 fold | 16
  2-<4 fold | 4
  4-<8 fold | 4
  >=8 fold | 12
  Missing | 3

ADVERSE EVENTS:
Time Frame: On treatment serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from start of study treament until the end of treatment visit for each participant (up to Week 180)
Description: On-treatment SAEs and non-serious AEs were reported for the Safety population consisted of all participants who received at least one dose of investigational product.
Arm/Group | Dolutegravir 50 mg BID
Serious Adverse Events (participants affected / at risk) | 46/183
Other Adverse Events (participants affected / at risk) | 143/183
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dolutegravir 50 mg BID (N=183)
Pneumonia (Infections and infestations) | 5
Progressive multifocal leukoencephalopathy (Infections and infestations) | 2
Pyrexia (General disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 3
Cytomegalovirus infection (Infections and infestations) | 1
Cytomegalovirus viraemia (Infections and infestations) | 1
Epstein-Barr virus infection (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Herpes ophthalmic (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Oesophageal candidiasis (Infections and infestations) | 1
Pneumococcal sepsis (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Streptococcal sepsis (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 2
Hepatic cirrhosis (Hepatobiliary disorders) | 1
Hepatitis acute (Hepatobiliary disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 1
Nerve compression (Nervous system disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Parotid gland enlargement (Gastrointestinal disorders) | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 2
Renal failure (Renal and urinary disorders) | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Immune reconstitution inflammatory syndrome (Immune system disorders) | 1
Alanine aminotransferase increased (Investigations) | 1
Ovarian mass (Reproductive system and breast disorders) | 1
Hypertensive emergency (Vascular disorders) | 1
Eye infection toxoplasmal (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Herpes virus infection (Infections and infestations) | 1
Bile duct obstruction (Hepatobiliary disorders) | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hodgkin's disease recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Syncope (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 2
Angina pectoris (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Bipolar disorder (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1
Hepatitis B (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 1
Orchitis (Infections and infestations) | 1
Anal cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lip and/or oral cavity cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Aphthous stomatitis (Gastrointestinal disorders) | 1
Hepatocellular injury (Hepatobiliary disorders) | 1
Nodular regenerative hyperplasia (Hepatobiliary disorders) | 1
Seizure (Nervous system disorders) | 1
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 1
Joint destruction (Musculoskeletal and connective tissue disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dolutegravir 50 mg BID (N=183)
Fatigue (General disorders) | 17
Pyrexia (General disorders) | 19
Asthenia (General disorders) | 13
Injection site reaction (General disorders) | 12
Diarrhoea (Gastrointestinal disorders) | 41
Nausea (Gastrointestinal disorders) | 26
Bronchitis (Infections and infestations) | 25
Upper respiratory tract infection (Infections and infestations) | 22
Nasopharyngitis (Infections and infestations) | 12
Rhinitis (Infections and infestations) | 11
Back pain (Musculoskeletal and connective tissue disorders) | 18
Arthralgia (Musculoskeletal and connective tissue disorders) | 12
Headache (Nervous system disorders) | 24
Cough (Respiratory, thoracic and mediastinal disorders) | 29
Rash (Skin and subcutaneous tissue disorders) | 17
Insomnia (Psychiatric disorders) | 14
Vomiting (Gastrointestinal disorders) | 13
Abdominal pain upper (Gastrointestinal disorders) | 14
Pruritus (Skin and subcutaneous tissue disorders) | 11
Constipation (Gastrointestinal disorders) | 12
Influenza (Infections and infestations) | 11
Sinusitis (Infections and infestations) | 11
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10
Anxiety (Psychiatric disorders) | 10
Hypertension (Vascular disorders) | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.